CLINICAL TRIAL: NCT03075761
Title: Physical Activity in Children at Risk of Post-thrombotic Sequelae: A Pilot Randomized Controlled Trial
Brief Title: Physical Activity in Children at Risk of Post-thrombotic Sequelae (PACT)
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Texas Scottish Rite Hospital for Children (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ayesha Zia, Assistant Professor of Pediatrics, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU 022016-057; 1K23HL132054-01 (NIH)
Record Dates: First submitted 2016-04-20; First posted 2017-03-09 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-03

CONDITIONS: Post Thrombotic Syndrome; Deep Vein Thrombosis
Keywords: Venous thromboembolism; Deep Vein Thrombosis; Lower Extremity; Blood clot; Anticoagulation; Physical Activity; Fitbit; Post-thrombotic syndrome; Post-phlebitic syndrome; Thrombosis
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis; Venous Thromboembolism; Thrombosis; Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants randomized to the intervention arm will receive a Fitbit, formal 30-minute education session on post-thrombotic syndrome (PTS) and benefits of increased physical activity. An individualized activity prescription will be provided and participants will be asked to maintain the target level of activity for 12 weeks after determining their habitual activity in the first 4 weeks.
  Interventions: Device: Fitbit; Behavioral: 30-minute education session
- Control (Active Comparator): Participants randomized to the control arm will receive a formal 30-minute education session on post-thrombotic syndrome (PTS) and the benefits of increased physical activity. Their physical activity will be self-reported in an activity log and by the Gordin activity questionnaire over the 16-week intervention period.
  Interventions: Behavioral: 30-minute education session

INTERVENTIONS:
Device: Fitbit — The Fitbit will be utilized in the intervention arm to improve adherence to a 12-week activity regimen.
  Other Names: Activity tracker
  Arms: Intervention
Behavioral: 30-minute education session

SUMMARY:
'The PACT trial' is randomized pilot trial to demonstrate the feasibility and potential effectiveness of a personal "fitness tracker" to improve adherence to an activity regimen following an initial acute DVT in children.

DETAILED DESCRIPTION:
The feasibility of an innovative intervention of a validated fitness tracker, the Fitbit, to improve adherence to a 12-week activity regimen in a pilot randomized controlled trial (RCT) will be tested in 44 subjects with first, acute, proximal lower extremity deep vein thrombosis (DVT).

The primary outcomes will consist of a) feasibility indicators determined a priori (eligibility, consent, adherence, retention) and b) estimates of effect size associated with the prescribed activity regimen, by describing within-subject change in QoL and potential biomarkers of postthrombotic syndrome (PTS) pre and post intervention in each group.

ELIGIBILITY:
Inclusion Criteria:

* A radiologically confirmed, acute, proximal first lower extremity DVT
* 4 to 8 weeks after starting anticoagulation
* Out-patient ambulatory status

Exclusion Criteria:

* Contraindication to increasing activity such as patients with juvenile arthritis, poor balance, congestive heart failure, etc.

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 111 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Zia, M.D, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hasan R, Hanna M, Zhang S, Malone K, Tong E, Salas N, Sarode R, Journeycake J, Zia A. Physical activity in children at risk of postthrombotic sequelae: a pilot randomized controlled trial. Blood Adv. 2020 Aug 11;4(15):3767-3775. doi: 10.1182/bloodadvances.2020002096. PMID 32780844

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 111 patients were screened, of whom 40 (36%) met study eligibility criteria. Of these, 23 (57.5%) consented to participate (11 randomized to physical activity arm and 12 to education or standard care arm)
Groups:
- Intervention: Participants randomized to the intervention arm will receive a Fitbit, formal 30-minute education session on post-thrombotic syndrome (PTS) and benefits of increased physical activity. An individualized activity prescription will be provided and participants will be asked to maintain the target level of activity for 12 weeks after determining their habitual activity in the first 4 weeks.
  Fitbit: The Fitbit will be utilized in the intervention arm to improve adherence to a 12-week activity regimen.
  30-minute education session
- Control: Participants randomized to the control arm will receive a formal 30-minute education session on post-thrombotic syndrome (PTS) and the benefits of increased physical activity. Their physical activity will be self-reported in an activity log and by the Gordin activity questionnaire over the 16-week intervention period.
  30-minute education session
Period: Overall Study
Arm/Group | Intervention | Control
Started | 11 | 12
Completed | 10 | 6
Not Completed | 1 | 6
Not completed — Lost to Follow-up | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.18 (2.04) | 14.25 (2.56) | 14.70 (2.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 10 | 8 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.83 (12.34) | 26.86 (5.58) | 28.28 (9.69)
OW/obese [Count of Participants; unit: Participants] — Participants were categorized to have normal weight if their BMI was between 5th and 85th, overweight for BMI between >85th-95th, and obese if BMI was ≥ 95th percentile for age and sex (Reference: Severe obesity in children and adolescents: identification, associated health risks, and treatment approaches: a scientific statement from the American Heart Association)
  Participants | 6 | 9 | 15
Clot burden at diagnosis occlusive [Count of Participants; unit: Participants] — Clot burden was defined as completely occlusive thrombus in at least one vein segment at VTE diagnosis.
  Participants | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Number of Participants Who Meet Study Eligibility Criteria at Baseline
Description: Feasibility criteria for rate of study eligibility met when assessed to be ≥ 30%
  INCLUSION CRITERIA:
  1.) Age 7-21 years 2.)2. A radiologically confirmed, acute, proximal (iliofemoral and femoropopliteal) first lower extremity DVT and/or confirmed, acute pulmonary embolism (unilateral or bilateral) 3.) 12 weeks (±2 weeks) after starting anticoagulation 4.) Out-patient ambulatory status
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Inpatients and Outpatients With VTE: All Inpatients and outpatients with VTE from following 3 sources:
  (1) new patient referrals to the Bleeding Disorders and Thrombosis outpatient clinic, (2) inpatient admissions to the hematology service, and (3) inpatient consultations for VTE that were not on primary hematology service.
Arm/Group | Inpatients and Outpatients With VTE
Number analyzed (Participants) | 111
Participants | 40

2. Primary Outcome: Number of Screened Subjects Who Provided Consent at Baseline
Description: Feasibility criteria for rate of consent was assessed to be ≥ 30% at baseline
  INCLUSION CRITERIA:
  1.) Age 7-21 years 2.)2. A radiologically confirmed, acute, proximal (iliofemoral and femoropopliteal) first lower extremity DVT and/or confirmed, acute pulmonary embolism (unilateral or bilateral) 3.) 12 weeks (±2 weeks) after starting anticoagulation 4.) Out-patient ambulatory status
Time Frame: Baseline
Population: For this specific outcome, we only assess the screened subjects who met the eligibility criteria are included in this cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Subjects Who Consented: Screened subjects who met the eligibility criteria are included in this cohort.
Arm/Group | Eligible Subjects Who Consented
Number analyzed (Participants) | 40
Participants | 23

3. Primary Outcome: Mean Number of Participants Who Adhered to the Assigned Physical Activity During 8-week Period (Intervention Arm -FitBit Arm )
Description: Adherence in the physical activity group is calculated based on the number of participants who complied with the target weekly goal or activity prescription during the "active" 8-week period.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: number of participants
Groups:
- FitBit Group's Adherence to Physical Activity: Targeted activity is defined as walking-jogging program to capture steps/day by the Fitbit during Active phase. If preferred or already involved, participants may perform strenuous muscle-strengthening or bone-strengthening exercises (eg, lifting weights, jumping rope, dancing, or team sports) to replace the walking-jogging program as long as the target goal for physical activity was met.
Arm/Group | FitBit Group's Adherence to Physical Activity
Number analyzed (Participants) | 11
number of participants | 3 (1.2)

4. Primary Outcome: Mean Physical Activity Questionnaire Score at 3 Months (Standard of Care Arm Only)
Description: The Godin-Shephard Leisure-Time Physical Activity Questionnaire was used to quantify physical activity levels. Individuals reporting moderate-to-strenuous activity levels ≥24 were classified as active (better outcome), whereas individuals reporting moderate-to-strenuous activity levels ≤23 were classified were insufficiently active (worse outcome).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Standard of Care Group's Adherence to Physical Activity: Proportion of participants who completed and submitted physical activity questionnaires.
Arm/Group | Standard of Care Group's Adherence to Physical Activity
Number analyzed (Participants) | 11
score on a scale | 56 (29)

5. Primary Outcome: Mean Physical Activity Questionnaire Score at 6 Months (Standard of Care Arm Only)
Description: as for outcome 4
Time Frame: 6 months
Population: Participants who submitted the questionnaire were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care Group's Adherence to Physical Activity
Number analyzed (Participants) | 10
score on a scale | 52 (32)

6. Primary Outcome: Mean Physical Activity Questionnaire Score at 9 Months (Standard of Care Arm Only)
Description: as for outcome 4
Time Frame: 9 months
Population: Participants who submitted the questionnaire were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care Group's Adherence to Physical Activity
Number analyzed (Participants) | 9
score on a scale | 38 (36)

7. Primary Outcome: Proportion of Subjects Who Complete Post-randomization
Description: Feasibility criteria is met when assessed to be ≥ 80%. This includes the number of subjects who successfully completed the trial.
Time Frame: Within 24 months of trial initiation
Population: For this specific outcome, we only assess the 11 subjects in the intervention arm and 12 subjects in the control arm.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Participants randomized to the intervention arm will receive a Fitbit, formal 30-minute education session on post-thrombotic syndrome (PTS) and benefits of increased physical activity. An individualized activity prescription will be provided and participants will be asked to maintain the target level of activity for 12 weeks after determining their habitual activity in the first 4 weeks.
  FitBit will be utilized in the intervention arm to improve adherence to a 12-week activity regimen.
  30-minute education session
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11 | 12
Participants | 10 | 6

8. Secondary Outcome: Change in PTS Biomarkers (D-dimer)
Description: Change in PTS biomarkers from baseline to post intervention of increased physical activity measured by coagulation activation marker D-dimer.
Time Frame: From baseline to 6 months
Population: For this specific outcome, we only assess the 11 subjects in the intervention arm and 12 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11 | 12
µg/mL | -4675 (5633) | -6241 (6780)

9. Secondary Outcome: Percentage Change From Baseline in FVIII PTS Biomarker
Description: Change in PTS biomarkers from baseline to post intervention of increased physical activity measured by the coagulation activation marker FVIII
Time Frame: From baseline to 6 month
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11 | 12
percent change | -39.6 (92) | -50.4 (82.5)

10. Secondary Outcome: Change in PTS Biomarkers (C-reactive Protein)
Description: Change in PTS biomarkers from baseline to post intervention of increased physical activity measured by inflammation marker C-reactive protein (CRP) using a latex-enhanced immunoturbidimetric assay.
Time Frame: From baseline to 6 month
Population: For this specific outcome, we only assess the 11 subjects in the intervention arm and 12 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11 | 12
mg/dL | -0.4 (1.6) | -0.6 (1.6)

11. Secondary Outcome: Change in PTS Biomarkers (Fibrinolysis - Endogenous Thrombin Potential)
Description: Change in PTS biomarkers from baseline to post intervention of increased physical activity measured by endogenous thrombin potential using calibrated automated thrombogram (CAT). CAT is a routine test that measures hyper- and hypocoagulability.
Time Frame: From baseline to 6 month
Population: For this specific outcome, we only assess the 11 subjects in the intervention arm and 12 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: nM*min
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11 | 12
nM*min | 41.0 (223) | -60.1 (148)

12. Secondary Outcome: Change in PTS Biomarkers (Fibrinolysis - Thrombin Generation)
Description: Change in PTS biomarkers from baseline to post intervention of increased physical activity measured by thrombin generation assay using calibrated automated thrombogram (CAT). CAT is a routine test that measures hyper- and hypocoagulability.
Time Frame: From baseline to 6 month
Population: For this specific outcome, we only assess the 11 subjects in the intervention arm and 12 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11 | 12
nmol/L | 60.5 (164) | 0.2 (28.4)

13. Secondary Outcome: Percent Change in Fibrinolysis Biomarker
Description: Percent Change in Fibrinolysis Biomarker from baseline to post intervention of increased physical activity is measured by thromboelastography (TEG). TEG is often used to predict bleeding and diagnose various bleeding disorders.
  Lysis 30% and Lysis 60% are measurements of percent amplitude reduction 30 and 60 minutes after maximum amplitude, respectively, on thromboelastography.
  Decreased clotting ability (negative value) = better outcome Increased clotting ability (positive value)= worse outcome
Time Frame: From baseline to 6 month
Population: For this specific outcome, we only assess the 11 subjects in the intervention arm and 12 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: percent amplitude change
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11 | 12
percent amplitude change
  Lysis 30, % (percent amplitude change 30 minutes after maximum amplitude) | -0.05 (3.3) | 2.1 (3.1)
  Lysis 60, % (percent amplitude change 60 minutes after maximum amplitude) | -0.04 (11.6) | 6.2 (6.5)

14. Secondary Outcome: Change in Quality of Life
Description: Change in Quality of Life from baseline to post intervention of increased physical activity assessed by PedsQL instrument. It consists of structured interview with the parents and the child with 23 items divided among 4 sub-scales to assess function in 4 domains: Physical; Emotional; social; and School. Each item is a statement of a problem, which the subject rates in severity from 0-4, indicating a problem never occurs (score of 0) to almost always occurs (score of 4). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50,3=25,4=0, with higher scores indicating better health related QoL.
  The positive change from baseline to 6 months correspond to better quality of life.
Time Frame: From baseline to 6 months
Population: For this specific outcome, we only assess the 11 subjects in the intervention arm and 12 subjects in the control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11 | 12
score on a scale | 5.4 (14.3) | 24.5 (14.2)

ADVERSE EVENTS:
Time Frame: From enrollment to end of treatment at 24 months
Description: Adverse events and serious adverse events were not collected as they were not the primary and secondary outcomes of the study.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT03075761/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT03075761/ICF_001.pdf